CLINICAL TRIAL: NCT02954874
Title: A Randomized, Phase III Trial to Evaluate the Efficacy and Safety of Pembrolizumab (MK-3475) as Adjuvant Therapy for Triple Receptor-Negative Breast Cancer With >/= 1 CM Residual Invasive Cancer or Positive Lymph Nodes (ypN1mi, ypN1-3) After Neoadjuvant Chemotherapy
Brief Title: Testing MK-3475 (Pembrolizumab) as Adjuvant Therapy for Triple Receptor-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01595; NCI-2016-01595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1418/BR006; s16-02231; S1418 (Other: SWOG); S1418 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Invasive Breast Carcinoma; Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Specimen Handling; Watchful Waiting; Observation; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (observation) (Experimental): Patients receive no treatment but are monitored at standard clinical intervals during first year after randomization. Patients are examined every 12 weeks for 1 year, every 6 months for 4 years, and then annually for 5 years. Patients may undergo radiation therapy within 12 weeks of last breast cancer operation or after treatment. Patients may also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Patient Observation; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on days 1 and 22. Cycles repeat every 42 days for 52 weeks in the absence of disease progression or unacceptable toxicity. Patients may undergo radiation therapy within 12 weeks of last breast cancer operation or after treatment. Patients may also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Patient Observation — Undergo standard monitoring
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm I (observation)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (pembrolizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This randomized phase III trial studies how well pembrolizumab works in treating patients with triple-negative breast cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare invasive disease-free survival (IDFS) of patients with triple-negative (TNBC) or low estrogen receptor (ER)-positive and/or HER2 borderline breast cancer who have >= 1 cm residual invasive breast cancer and/or positive lymph nodes (ypN1mi, ypN1, ypN2, ypN3) after neoadjuvant chemotherapy randomized to receive 1 year of MK-3475 (pembrolizumab) adjuvant therapy compared to no MK-3475 (pembrolizumab), in both the entire study population and also in the PD-L1 positive subset.

SECONDARY OBJECTIVES:

I. To compare the effects of MK-3475 (pembrolizumab) on overall survival (OS) and distant recurrence-free survival (DRFS) between the two randomized arms for the PD-L1 positive patients and then all patients.

II. To assess the toxicity and tolerability of MK-3475 (pembrolizumab) in this patient population with or without radiation therapy.

BEHAVIORAL AND HEALTH OUTCOMES (BAHO) STUDY OBJECTIVES:

I. To examine the association between biomarkers of inflammation and quality of life and patient reported outcomes between the two groups during and at the end of therapy.

II. To examine the long-term and late effects of treatment on patient-reported outcomes.

ADDITIONAL OBJECTIVE:

I. To collect tissue and whole blood for processing and banking in anticipation of future correlative studies in this patient population.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (OBSERVATION): Patients receive no treatment but are monitored at standard clinical intervals during first year after randomization. Patients are examined every 12 weeks for 1 year, and every 6 months for 4 years, then annually for 5 years.

ARM II (PEMBROLIZUMAB): Patients receive pembrolizumab intravenously (IV) over 30 minutes on days 1 and 22. Cycles repeat every 42 days for 52 weeks in the absence of disease progression or unacceptable toxicity.

All patients may undergo radiation therapy within 12 weeks of last breast cancer operation or after treatment. Patients may also undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for 5 years, then annually thereafter until 10 years from treatment randomization.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION
* Patients must have histologically confirmed estrogen receptor (ER)-, progesterone receptor (PR)- and HER2-negative (triple-negative, TNBC) or ER-, PR- weakly positive and/or HER2- equivocal status and must not have received and not be planning to receive adjuvant anti-HER2 or endocrine therapies after completion of neoadjuvant chemotherapy; patients who are HER2-positive by American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines are ineligible; HER2-negative and HER2-equivocal cases as per ASCO CAP guidelines that do not receive HER2-targeted therapy are eligible; patients with weakly ER or PR positive disease, defined as ER and/or PR less than or equal to (=<) 5% by immunohistochemistry, are eligible if the treating physician considers the patient not eligible for adjuvant endocrine therapy; residual disease must be >= 1 cm in greatest dimension, and/or have positive lymph nodes (ypN1mi, ypN1, ypN2, ypN3) observed on pathologic exam

  * NOTE: If the ER and/or HER2 results are discordant between the initial, pre-chemotherapy, and post-chemotherapy surgical tissue, the receptor status of the residual disease has to be used to determine eligibility. Immunohistochemistry (IHC)-positive isolated tumor cells in the lymph node (N0 [i+]) are not considered node-positive and these patients also must have >= 1 cm residual invasive cancer in the breast to be eligible.
* Patients must not have metastatic disease (i.e., must be clinically M0 or Mx; systemic staging studies with imaging should follow routine practice as per National Comprehensive Cancer Network [NCCN] and ASCO guidelines); patients must not have locally recurrent disease
* It is preferred that axillary lymph node sampling is performed after completion of neoadjuvant chemotherapy to allow more accurate assessment of pathologic response; complete axillary lymph node dissection (ALND) after neoadjuvant chemotherapy is recommended in the following situations:

  * Patients had documented pathologic involvement of the axillary nodes (fine needle aspiration [FNA] or core biopsy) before neoadjuvant chemotherapy and had sentinel node biopsy after neoadjuvant chemotherapy with positive sentinel node(s)
  * Patient had documented pathologic involvement of the axillary nodes (FNA or core biopsy) before neoadjuvant chemotherapy and had only 1 sentinel lymph node removed after neoadjuvant chemotherapy

    * Except for (i) patients participating in the Alliance A11202 trial) or (ii) if the treating surgeon determines that a complete ALND is not in the best interest of the patient
    * NOTE: Patients who undergo sentinel node biopsy before starting neoadjuvant treatment and do not undergo post neoadjuvant assessment of the axillary nodes or who have negative axillary nodes on post neoadjuvant assessment must have >= 1 cm residual invasive cancer in the breast after completion of neoadjuvant chemotherapy
* Patients must have a minimum of five, available unstained formalin-fixed paraffin-embedded (FFPE) slides (4-5 micron thickness) from the residual (post-neoadjuvant) invasive tumor in primary site or lymph node; (these will be submitted to a central laboratory to determine PD-L1 expression); the tumor tissue must be adequate for PD-L1 testing, which typically requires a minimum of 100 cancer cells per slide; local PD-L1 results, even if available, will not substitute for central testing

  * NOTE: Initial order for specimen kits should be placed at least two weeks prior to registering the first patient at each site
* Patients must be offered the opportunity to participate in specimen banking
* The BAHO substudy was permanently closed to accrual on June 23, 2020, and willingness of English-speaking patients to participate in the BAHO substudy is no longer applicable
* Patients must have had neoadjuvant chemotherapy followed by surgery; the choice of neoadjuvant chemotherapy is determined by the treating physician; we recommend following the National Comprehensive Cancer Network (NCCN) treatment guidelines for TNBC; patients who cannot complete all planned treatment cycles for any reason are considered high risk and therefore are eligible for the study if they have residual disease; patients must have resolution of adverse event(s) of the most recent prior chemotherapy to grade 1 or less, except alopecia and =< grade 2 neuropathy which are allowed
* Patients may receive post-operative (adjuvant) chemotherapy for up to 24 weeks of duration (e.g. 8 cycles of capecitabine as in the Capecitabine for Residual Cancer as Adjuvant Therapy (CREATE-X) trial; the 24-week duration does not include treatment delays) after completion of surgery at the discretion of the treating physician; co-enrollment to EA1131 is allowed, provided that patients complete or discontinue adjuvant chemotherapy prior to step 1 registration; at the time of step 1 registration, patients must have resolution of adverse event(s) of the most recent prior chemotherapy to =< grade 1, except alopecia and =< grade 2 neuropathy which are allowed; patients that have received adjuvant chemotherapy (including via co-enrollment to EA1131) must be registered to step 1 within 35 days after final dose of adjuvant chemotherapy
* Patients must have completed their final breast surgery (rendering them free from disease) with clear resection margins for invasive cancer and DCIS within the following timelines:

  * 90 days prior to step 1 screening registration for patients not receiving post-operative (adjuvant) chemotherapy OR
  * 270 days prior to step 1 screening registration for patients who have received post-operative (adjuvant) chemotherapy Positive margins are allowed only if the surgical team of the patient deems further resection impossible
* Patients for whom radiation therapy (RT) to the affected breast or chest wall and regional nodal areas is clinically indicated as per NCCN treatment guidelines, should receive routine RT after randomization when possible, and receive MK-3475 (pembrolizumab) concurrent with RT, if randomized to the experimental arm; however, routine RT administered, or initiated, prior to registration is also allowed; MK-3475 (pembrolizumab) may be added to ongoing radiation, or started after its completion, if randomized to the experimental arm, provided there are no > grade 1 radiation-related skin toxicities and provided that no radiosensitizing chemotherapy is being administered; co-enrollment in the Alliance A221505 (NCT03414970) and A011202 (NCT01901094) trials or in the NSABP-B51 (NCT01872975) trial is allowed, but patients must not be planning to receive radiation therapy given on these trials concurrently with MK-3475 (pembrolizumab) treatment on S1418/BR006; whether or not patient will receive RT and the extent of intended RT must be specified at time of registration; NOTE: Patients who receive post-operative chemotherapy may receive radiation therapy before or after the chemotherapy; a short course of reduced dose chemotherapy or other agents concomitant with radiation for radiation sensitization is not considered to be adjuvant chemotherapy
* Patients must not have had prior immunotherapy with anti-PD-L1, anti-PD-1, anti-CTLA4 or similar drugs; patients must not be planning to receive any of the prohibited therapies during the screening or treatment phases of the study
* Patients must not be planning to receive concomitantly other biologic therapy, hormonal therapy, other chemotherapy, surgery or other anti-cancer therapy except radiation therapy while receiving treatment on this protocol; however, patients receiving extended adjuvant endocrine therapy for an earlier ER positive breast cancer treated with curative intent and without recurrence for at least 5 years may continue with their endocrine therapy; elective surgery or surgery that is not related to cancer therapy is allowed, at the discretion of the treating investigator
* Patients must be >= 18 years of age
* Patients must have Zubrod performance status =< 2
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or evidence of active pneumonitis within 2 years prior to registration
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine for pre-existing hypothyroidism, insulin for type I diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients must not have received live vaccines within 30 days prior to registration; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to registration; patients who have completed curative therapy for HCV are eligible; patients with known human immunodeficiency virus (HIV) infection are eligible if they meet each of the following 3 criteria:

  * CD4 counts >= 350 mm^3
  * Serum HIV viral load of < 25,000 IU/ml and
  * Treated on a stable antiretroviral regimen
* No other prior invasive malignancy is allowed except for the following: adequately treated basal (or squamous cell) skin cancer, in situ breast or cervical cancer; stage I or II invasive cancer treated with a curative intent without evidence of disease recurrence for at least five years
* Patients must have complete history and physical examination within 28 days prior to registration
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent for this protocol in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2 REGISTRATION
* Patients must not be registered to step 2 until receiving confirmation from the Southwest Oncology Group (SWOG) Statistical and Data Management Center that the patient's tissue specimen was adequate for PD-L1 testing; patients must be registered within 14 days of receiving the e-mail notification confirming submission was evaluable for PD-L1 status
* Absolute neutrophil count (ANC) >= 1,500 microliter (mcL) (obtained within 28 days prior to step 2 registration)
* Platelets >= 100,000/mcL (obtained within 28 days prior to step 2 registration)
* Hemoglobin >= 9 g/dL (obtained within 28 days prior to step 2 registration)
* A serum thyroid-stimulating hormone (TSH) and/or free T4 must be obtained within 28 days prior to step 2 registration to obtain a baseline value
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) (obtained within 28 days prior to step 2 registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x IULN (obtained within 28 days prior to step 2 registration)
* Alkaline phosphatase =< 2.5 x IULN (obtained within 28 days prior to step 2 registration)
* Serum creatinine =< IULN OR measured or calculated creatinine clearance >= 60 mL/min (obtained within 28 days prior to step 2 registration)
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 day prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or vasectomy; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures; patients must not be pregnant or nursing; women of childbearing potential must plan to have a urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required
* Patients must not have an active infection requiring systemic therapy at the time of starting therapy
* Site must verify that there is no known change in the step 1 eligibility since initial registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1155 (Estimated)
Dates: Start 2017-01-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | From date of randomization to date of first invasive recurrence, second invasive primary cancer (breast or not), or death due to any cause, assessed up to 10 years
  The distributions of IDFS will be estimated using the Kaplan-Meier method, with 95% confidence intervals (CI) calculated using Greenwood's formula. Comparisons between the two treatment arms will be performed using the stratified log-rank test. The hazard ratios and 95% CIs will be based on the stratified Cox proportional hazard model with treatment as the only covariate. Secondary analyses of IDFS will be performed to describe consistency or divergence across subgroups. This will include a forest plot of treatment hazard ratios and associated 95% confidence intervals for each level of the stratification factors and major prognostic covariates (such as use of radiation therapy). The statistical significance of the interaction between treatment and each stratification factor or prognostic variable will be assessed.
Severity of fatigue | 55 weeks after randomization
  Measured by Patient Reported Outcomes Measurement Information System (PROMIS) fatigue scale. Will be compared between the two treatment groups by means of multiple linear regression with adjustment for the corresponding baseline measurement as well as whether or not the patient received radiation therapy which is known to be associated with post-treatment fatigue. No multiple comparisons adjustment will be employed since these outcomes evaluate the toxicity of the investigational drug. The clinical meaningfulness of each comparison will be considered.
Physical function | 55 weeks after randomization
  Reported by patients measured by PROMIS Global physical health scale. Will be compared between the two treatment groups by means of multiple linear regression with adjustment for the corresponding baseline measurement as well as whether or not the patient received radiation therapy which is known to be associated with post-treatment fatigue. No multiple comparisons adjustment will be employed since these outcomes evaluate the toxicity of the investigational drug. The clinical meaningfulness of each comparison will be considered.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 10 years
  The distributions of OS will be estimated using the Kaplan-Meier method, with 95% CI calculated using Greenwood's formula. Comparisons between the two treatment arms will be performed using the stratified log-rank test. The hazard ratios and 95% CIs will be based on the stratified Cox proportional hazard model with treatment as the only covariate.
Distant recurrence-free survival (DRFS) | From date of randomization to date of invasive distant disease recurrence, second invasive primary cancer (breast or not) or death due to any cause, assessed up to 10 years
  The distributions of DRFS will be estimated using the Kaplan-Meier method, with 95% CI calculated using Greenwood's formula. Comparisons between the two treatment arms will be performed using the stratified log-rank test. The hazard ratios and 95% CIs will be based on the stratified Cox proportional hazard model with treatment as the only covariate.
Incidence of adverse events | Up to 10 years
  Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Toxicity analysis will be conducted in all patients receiving at least one dose of MK-3475 (pembrolizumab). The incidence of adverse events will be reported.
Severity and frequency of treatment-related symptoms (diarrhea, nausea, rash, cough, and shortness of breath, musculoskeletal pain) over time of patients receiving pembrolizumab | Up to 10 years
  Compared without treatment. The distributions of the corresponding Patient Reported Outcomes version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) items will be compared between the two treatment groups using a mixed ordinal logistic regression model for repeated measures. The model will also include the corresponding baseline measurement and time. Presence of treatment-by-time interaction will be tested for each of these endpoints. Similar analyses will be performed for disease related symptoms. The descriptive and graphical methods suggested in Basch, et. al. will be used to summarize the distributions of different symptoms by treatment group over time.
Emotional function and disease-related symptoms in patients receiving pembrolizumab | Up to 10 years
  Assessed by PROMIS global mental health scale score. Will be compared between the two treatment groups using a mixed model for repeated measures analysis with adjustment for the baseline score and time. Presence of treatment-by-time interaction will be investigated.
Impact of treatment and treatment-related symptoms on physical function in patients without therapy | 55 weeks after randomization
  Compared to patients receiving pembrolizumab. A multiple linear regression model will be performed with physical health scale score as an outcome and treatment and treatment related symptoms as covariates. Presence of treatment by each individual symptom item interactions will be investigated.
Relationship between treatment-related symptoms and adherence to the study medication | Up to 10 years
  Will be investigated among patients randomized to pembrolizumab treatment group by means of multiple logistic regression. Patients who have been on study therapy for 70% or more of their expected time on therapy will be considered adherent.
Resolution of treatment-related symptoms in patients receiving pembrolizumab | 18 months after randomization
  Compared to patients without treatment. A change in severity of the particular symptom will be compared between the two treatment groups by means of multiple linear regression with adjustment for the corresponding measurement at the 55 week assessment point.
Long-term quality of life and symptoms between the two treatment groups | Up to 60 months after randomization
  Mixed models for repeated measures analysis will be used with adjustment for scores at 18 months to examine changes in physical and emotional domain scores, fatigue and other persistent symptoms over the course
Role of pro-inflammatory cytokines in the development of pembrolizumab associated symptoms | Up to 55 weeks
  Specifically focused on treatment-associated fatigue. This will be compared to patients in the observation group.
Single nucleotide polymorphisms (SNPs) in the promotor region of pro-inflammatory cytokine genes and the risk for development and severity of treatment-associated fatigue and other symptoms | Up to 10 years
  The role of these SNPs in the persistence of long-term fatigue in all patients will also be explored using treatment assignment as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, Principal Investigator — SWOG Cancer Research Network
Locations (920):
- United States (896):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern Cancer Center PC-Daphne, Daphne, Alabama
  - Southern Cancer Center PC-Mobile, Mobile, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Southern Cancer Center PC-Springhill, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Community Cancer Institute, Clovis, California
  - City of Hope Corona, Corona, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - City of Hope Mission Hills, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Huntington Memorial Hospital, Pasadena, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Mac Neal Hospital, Berwyn, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - MercyOne Genesis Silvis Cancer Center, Silvis, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - CHRISTUS Saint Patrick Hospital, Lake Charles, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - New England Cancer Specialists - Kennebunk, Kennebunk, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - New England Cancer Specialists - Topsham, Topsham, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - York Hospital, York Village, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Michigan State University, East Lansing, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Covenant Health Cancer Centers, Knoxville, Tennessee
  - Covenant Health Cancer Centers - West, Knoxville, Tennessee
  - Covenant Health Oncology Group - Lenoir City, Lenoir City, Tennessee
  - Covenant Health Oncology Group - Maryville, Maryville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Covenant Health Oncology Group - Oak Ridge, Oak Ridge, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Austin Cancer Centers-Central Austin, Austin, Texas
  - Houston Methodist San Jacinto Hospital, Baytown, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
- Canada (20):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHU de Quebec-Hopital du Saint-Sacrement (HSS), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Puerto Rico (4):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - San Juan City Hospital, San Juan